CLINICAL TRIAL: NCT04770428
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Multiple Doses of MEDI7352 Administered by the Subcutaneous Route in Healthy Japanese and Caucasian Subjects
Brief Title: Evaluate Safety, Tolerability, Pharmacokinetics and Immunogenicity of MEDI7352 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5680C00004; 2020-005982-14 (EudraCT Number)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Painful Osteoarthritis of the Knee
Keywords: MEDI7352; Bi-specific fusion protein; Multiple doses; Subcutaneous route; Pharmacokinetics; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is double-blinded with regard to treatment (MEDI7352 or placebo) for all placebo-controlled dose groups (groups where placebo and active substance is given in a cohort, ie, the Sponsor, the Investigator, all clinical staff involved in the clinical study, the participants, and the study monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Japanese MEDI7352 (Experimental): Randomized Japanese participants will receive single doses of MEDI7352 subcutaneously.
  Interventions: Drug: MEDI7352
- Cohort 1: Japanese Placebo (Placebo Comparator): Randomized Japanese participants will receive matching placebo subcutaneously.
  Interventions: Drug: Placebo
- Cohort 2: Caucasian MEDI7352 (Experimental): Randomized Caucasian participants will receive single doses of MEDI7352 subcutaneously.
  Interventions: Drug: MEDI7352
- Cohort 2: Caucasian Placebo (Placebo Comparator): Randomized Caucasian participants will receive matching placebo subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI7352 — A dose of MEDI7352 will be administered as two 1.5 mL injections in the abdomen. Following an overnight fast of at least 8 hours, each participant will receive a single dose of MEDI7352 on 4 occasions.
  Arms: Cohort 1: Japanese MEDI7352; Cohort 2: Caucasian MEDI7352
Drug: Placebo — Matching placebo will be administered as two 1.5 mL injections in the abdomen. To maintain the double-blind requirements, the placebo volume administered will be equivalent to the MEDI7352 volume administered for each dosing. Following an overnight fast of at least 8 hours, each participant will receive matching placebo on 4 occasions.
  Arms: Cohort 1: Japanese Placebo; Cohort 2: Caucasian Placebo

SUMMARY:
This study will evaluate safety, tolerability, pharmacokinetics and immunogenicity of MEDI7352 in healthy participants.

DETAILED DESCRIPTION:
The study will comprise:

* A Screening Period of up to 36 days (approximately 5 weeks);
* A Treatment Period of 6 weeks where participants will be given 1 dose of study treatment every 2 weeks (4 doses in total). Participants will be required to stay in the Clinical Unit from Days -1 to 8 (Visit 2), from Days 14 to 15 (Visit 6), from Days 28 to 29 (Visit 9), and from Days 42 to 50 (Visit 12). In addition, participants will have multiple visits to the Clinical Unit to complete the study assessments;
* A Follow-up Period of 42 days (6 weeks) where participants will also have multiple visits to the Clinical Unit to complete the study assessments, and;
* A final Follow-up Visit after 42 days after the Treatment Period.

Participants will receive fixed multiple subcutaneous (SC) doses of MEDI7352 or placebo on 4 occasions; one dose every 2 weeks on Days 1, 15, 29 and 43, under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female of non childbearing potential participants aged 18 to 65 (inclusive) years for Caucasian participants and 20 to 65 (inclusive) years for Japanese participants with suitable veins for cannulation or repeated venepuncture
* Japanese or Caucasian ethnicity
* Post-menopausal women must have had ≥ 12 months of spontaneous amenorrhea with an follicle stimulating hormone (FSH) concentration consistently ≥ 40 mIU/mL and a negative serum or urine pregnancy test result at Screening or Day -1. Surgically sterile women must have had a hysterectomy, and bilateral ovariectomy (oophorectomy), must provide documentation of the procedure and have had a negative serum or urine pregnancy test at Screening or Day -1. An intermediate or positive pregnancy test, can be confirmed by repeating the pregnancy test and demonstrating non-doubling of β-human chorionic gonadotropin levels every 48 to 72 hours
* Men who are biologically capable of fathering children must agree and commit to use of an adequate form of a highly effective method of contraception and refrain from sperm donation for the duration of the Treatment Period and for 3 months after the last administration of study treatment
* Body mass index 18 and 30 kg/m^2, weight at least 50 kg
* No clinically significant abnormality identified on medical or laboratory evaluation at Screening unless the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures
* 12-lead electrocardiogram recorded at Screening and Day -1 that is normal for the age group and shows no significant abnormalities that will compromise safety
* Physical examinations with no significant findings at Screening and on Day -1.

Exclusion Criteria:

* Participation in another clinical study or use of any experimental medication, device, or biologic with an investigational product (IP) within 5 half-lives of that IP or 3 months (whichever is longer) prior to first dosing
* Participation in another study investigating any form of anti-NGF or anti-TNF therapy in the 6 months prior to Screening and until after the final Follow-up Visit
* Any positive laboratory result at screening for COVID-19
* Blood donation or draw in excess of 400 mL within 2 months prior to Screening or plasma donation in excess of 50 mL within 30 prior to Screening
* Inability to comply with study-related restrictions and requirements related to consumption of alcohol, provision of meals and snacks, nicotine use, activity, blood donation, and contraception
* History of severe allergy/hypersensitivity reactions or ongoing severe allergy/hypersensitivity reactions, or history of hypersensitivity to immunizations or immunoglobulins or other biological modalities
* History of any significant psychiatric disorder
* Any clinically significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal, metabolic, GI, urologic, immunologic, rheumatologic or endocrine disease or disorder
* Recent (within the last 3 months) or active infection considered to be clinically significant, or any infection for which there are unresolved medical sequelae
* Clinically significant osteoarthritis (OA) currently affecting a major joint in the upper or lower extremity or axial spine; or other degenerative disease affecting any joint in participants for whom, there is an identified risk of osteonecrosis, rapidly progressing OA, subchondral insufficiency fractures, neurogenic arthropathy, or analgesia-induced arthropathy; or history of trauma or surgery involving any major joint or axial spine
* Radiological significant abnormalities reported on baseline MRI of hips and knees that are considered to present a risk of osteonecrosis, rapidly progressive OA, subchondral insufficiency fractures; or other coincidental finding(s) that present a risk to the safety or welfare of the participant
* History of excessive alcohol intake
* History of cancer within 5 years, with the exception of non-metastatic basal cell carcinoma of the skin, carcinoma in situ of the cervix or non-progressive prostate cancer
* History of drug abuse or positive test for drugs of abuse or alcohol
* Use of prescription or non-prescription drugs, including vitamins and herbal and dietary supplements, within 7 days or 5 half-lives of the drug (whichever is longer) prior to the administration of study treatment
* Any clinically important or significant abnormality on a physical examination, vital signs, ECG or clinical laboratory test results that could be detrimental to participant safety or compromise the study
* Positive serologic findings at Screening for Human immunodeficiency virus antibodies, hepatitis B surface antigen or hepatitis C virus antibodies
* Positive QuantiFERON test for tuberculosis
* Any minor medical or surgical procedure or trauma within 28 days of Day 1 or planned surgical procedure during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Upto Final Follow-up (Day 84) or Early Termination
  To evaluate the safety and tolerability of MEDI7352 in healthy Japanese and Caucasian participants following multiple dosing by the SC route

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to pharmacokinetic (PK) following multiple dosing by the SC route.
Time of Cmax (tmax) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Area under the serum concentration-time curve from time 0 to infinity (AUCinf) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Area under the serum concentration-time curve from time 0 to the time of the last quantifiable serum concentration (AUClast) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Area under the serum concentration-time curve for the dosing interval (AUCτ) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Average drug concentration over a dosing interval (Cavg) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Apparent volume of distribution at steady state (Vss/F) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Half-life (t1/2) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Apparent total body clearance (CL/F) for MEDI7352 | 1st dose: pre-dose (Day 1), post-dose Day 2, 4, 6, 8, 10 and 12; 2nd and 3rd doses: pre-dose (Days 15 and 29) and 7 days post-dose (Days 22 and 36); 4th dose: pre-dose (Day 43), post-dose Days 44, 46, 48, 50, 52, 54, 57, 64, 71
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to PK following multiple dosing by the SC route.
Number of participants with positive/negative antidrug antibodies (ADA) result for MEDI7352 | Days 1, 15, 29 and 43 and at Follow-up Visit (Days 50, 64, and 84)
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to immunogenicity following multiple dosing by the SC route.
ADA titers testing for all ADA-positive samples as measure of immunogenicity | Days 1, 15, 29 and 43 and at Follow-up Visit (Days 50, 64, and 84)
  To further assess MEDI7352 in healthy Japanese and Caucasian participants with respect to immunogenicity following multiple dosing by the SC route.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home